CLINICAL TRIAL: NCT01155427
Title: A Systematic Review of Literature on Common Antiretroviral Treatments Against Hepatitis B Virus (HBV)
Brief Title: Systematic Review of Antiretroviral Treatments for Chronic Hepatitis B (CHB)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Bristol-Myers Squibb, Study Director
Other Study IDs: AI463-186
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- entecavir: Patients initiating special antiviral treatments for CHB
- tenofovir: Patients initiating special antiviral treatments for CHB
- lamivudine: Patients initiating special antiviral treatments for CHB
- telbivudine: Patients initiating special antiviral treatments for CHB
- adefovir: Patients initiating special antiviral treatments for CHB

SUMMARY:
The purpose of this study is to support the clinical value of entecavir by assessing the relationship between viral load and histological improvement.

DETAILED DESCRIPTION:
Systematic review of prospective clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Patients with CHB diagnosis and no co-infection with Hep A, Hep C, Hep D, or HIV
* Age 16 years or older
* No post-transplant patients
* RCT, non-randomized trials, prospective cohort studies, prospectively analyses case series published since 2003
* At least one arm of trial must include monotherapy with entecavir, lamivudine, tenofovir, adefovir, or telbivudine
* Study arms must include at least 10 patients
* Follow-up of at least 48 weeks
* Published results available in English language

Exclusion Criteria:

* N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical trial enrollees
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Viral load
Histological improvement

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm